CLINICAL TRIAL: NCT00454597
Title: PHASE 1 The Effect of the Omentectomy on the Hyperglycemia and the Resistance to the Insulin in Patients With Morbid Obesity
Brief Title: Effect of the Omentectomy on the Hyperglycemia and the Resistance to the Insulin in Patients With Morbid Obesity
Acronym: omentectomy
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Universidad de Guanajuato (Other)
Responsible Party: arturo reyes hernandez, universidad de guanajuato
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 0910-0459; ID :0910-0459
Record Dates: First submitted 2007-03-27; First posted 2007-04-02 (Estimated); Last update posted 2008-06-04 (Estimated); Status verified 2008-05

CONDITIONS: Obesity; Diabetes Mellitus Type 2
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: omentectomy — surgery omentectomy

SUMMARY:
To determine if the omentectomy diminishes hyperglycemia and improves the resistance to the insulin in patients with morbid obesity and propensity to develop to Diabetes Mellitus type 2.

DETAILED DESCRIPTION:
To determine the Blood levels of glucose, curve of tolerance to the glucose, hemoglobin glycosylated, insulin, triglyceride, cholesterol, HDL, LDL, leptin and Adiponectin in patients with Obesity Morbid and that will be put under umbilical surgery and cholecystectomy opened.

To put under them umbilical surgery or Cholecystectomy open with and without omentectomy To compare the Blood levels of of glucose, curve of tolerance wing glucose, hemoglobin glycosylated, insulin, triglyceride, cholesterol, HDL, LDL, leptin and Adiponectin before and after the procedure

ELIGIBILITY:
Inclusion Criteria:

* All the patients with Obesity Morbid who suffer of hernia umbilical Chronic Cholecystitis Lithiasic non worsened.
* Patient with age between the 18 to 55 years of age.
* Both sorts.
* Patient with index of corporal mass from 30 to 35.
* Patient with index waist greater or equal hip of 100cm in men and women greater of 88cm.
* Patient that has a central glucose of 100 to 125mg.
* Patient that has a tolerance to the glucose of 140 to 200mg.
* Patient which they have a result of triglyceride in blood of 300 or greater.
* Patient that has values of LHD below 40 mg/dl.

Exclusion Criteria:

* Patient that they have I diagnose already established of Diabetes Mellitus type 2 and in medical treatment.
* Patient with elevation of hepátic enzymes (more than 50% of the superior limits of normality) and/or creatinin in 1,5 serum > mg/Dl.
* Patient with Diabetic ketoacidosis history.
* Uso of oral anticoagulants.
* Positive Test of pregnancy (Human Chorionic Gonadotropin ) for women.
* Recurrent Infections and at the time of the study.
* Umbilical Hernia complicated and strangled or Worsened Chronic Cholecystitis.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2007-02; Primary Completion 2007-03 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
To compare the Blood levels of of glucose, curve of tolerance wing glucose, hemoglobin glycosylated, insulin, triglyceride, cholesterol, HDL, LDL, leptin and Adiponectin before and after the procedure | 3 months

SECONDARY OUTCOMES:
To evaluate the metabolic conditions of the subjects of both groups to the 15 days and the month, 6, 12 and 24 months later to the procedure | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Arturo MD Reyes Hernandez, Surgery, Principal Investigator — Universidad de Guanajuato, Facultad de Medicina de León, Hospital General Regional de León
Locations (1):
- Hospital General Regional de León, Universidad de Guanajuato, Facultad de Medicina de León, León, Guanajuato, Mexico

REFERENCES:
- [Result] Thorne A, Lonnqvist F, Apelman J, Hellers G, Arner P. A pilot study of long-term effects of a novel obesity treatment: omentectomy in connection with adjustable gastric banding. Int J Obes Relat Metab Disord. 2002 Feb;26(2):193-9. doi: 10.1038/sj.ijo.0801871. PMID 11850750